CLINICAL TRIAL: NCT06920147
Title: PRevention Of Trauma-related Infections Through an Embedded Clinical Trials (PROTECT) Network
Brief Title: PRevention Of Trauma-related Infections Through an Embedded Clinical Trials Network
Acronym: PROTECT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Surgical Infection Society (Unknown)
Responsible Party: Principal Investigator, Lillian Kao, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-MS-24-0212
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ertapenem; Cefazolin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ertapenem only (Experimental)
  Interventions: Drug: Ertapenem
- Combination of cefazolin and metronidazole. (Experimental)
  Interventions: Drug: Cefazolin and Metronidazole.

INTERVENTIONS:
Drug: Ertapenem — Participants will receive a single dose of IV ertapenem (1g) in the operating room prior to incision or as soon as possible given the patient's hemodynamic status
  Arms: Ertapenem only
Drug: Cefazolin and Metronidazole. — Participants will receive a single dose of a combination of IV cefazolin (re-dosed during the case every 4 hours and/or after every 1,500 mL of blood loss) and IV metronidazole (single dose 500 mg) in the operating room prior to incision or as soon as possible given the patient's hemodynamic status
  Arms: Combination of cefazolin and metronidazole.

SUMMARY:
The purpose of this study is to compare the effectiveness of 2 prophylactic antibiotic regimens, ertapenem and cefazolin with metronidazole, in preventing organ space surgical site infections (OS-SSI) after emergency trauma laparotomy embedded into routine clinical care and to validate a Bayesian OS-SSI risk calculator using Trauma Quality Improvement Program (TQIP) standardized variables

ELIGIBILITY:
Inclusion Criteria:

* Trauma laparotomy within 90 minutes of arrival

Exclusion Criteria:

* Patients with a known allergy to cephalosporins or β-lactamase inhibitors
* Prisoners
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have post-laparotomy OS-SSIs | 30 days after surgery

SECONDARY OUTCOMES:
Number of participants that have superficial incisional SSIs | 30 days after surgery
Number of participants that have deep incisional SSIs | 30 days after surgery
Number of patients that show highest Clavien-Dindo grade for OS-SSIs | 30 days after surgery
  grades range from I (minor, requiring no intervention) to V (death)
Number of unplanned reoperations | 30 days after surgery
Number of readmissions | 30 days after surgery
Number of participants that have Clostridium difficile infections | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No